CLINICAL TRIAL: NCT02858856
Title: Sipjeondaebo-tang for Alleviating Fatigue Measured by Brief Fatigue Inventory and EORTC-QLQ-C30, BR23 Score Change Among Patients With Breast Carcinoma Receiving Chemotherapy
Brief Title: Clinical Trial of Sipjeondaebo-tang on Fatigue of Breast Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyunghee University Medical Center (Other)
Collaborators: Catholic Kwandong University (Other)
Responsible Party: Principal Investigator, Seong-Gyu Ko, Prof., Kyunghee University Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: ISEE_2016_SJDBT
Record Dates: First submitted 2016-07-30; First posted 2016-08-08 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — juzentaihoto

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A group (Experimental): Take Sipjeondaebo-tang on 0~2 week, 3~5 week of clinical trial period, total of 4 weeks
  Interventions: Drug: Sipjeondaebo-tang
- B group (Experimental): Take Sipjeondaebo-tang on 6~8 week, 9~11 week of clinical trial period, total of 4 weeks
  Interventions: Drug: Sipjeondaebo-tang

INTERVENTIONS:
Drug: Sipjeondaebo-tang — Herbal medicine which is a compound of 10 herbs.
  Other Names: Deciten granule

SUMMARY:
This is a pilot study that investigate efficacy and safety of Sipjeondaebo-tang on fatigue of patients with breast carcinoma receiving chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* men and women aged over 18 years
* patients who have histologically or cytologically confirmed breast tumor
* patients who applicable AC(doxorubicin + cyclophosphamide)
* ECOG score 0 to 2

Exclusion Criteria:

* patient impossible to orally intake
* patient with dementia, delirium and depression
* patient suffering from diseases like chronic hepatitis B, C or hepatocirrhosis
* severe liver disability (3-fold the normal high range value for ALT, AST)
* patient who has diabetes not controlled by diet, hypertension, hyperthyroidism,
* severe systemic disease
* use of other investigational products within the past 30 days
* hypersensitivity to investigational product
* others who are judged not to be appropriate to study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2017-03-20 (Actual); Primary Completion 2018-03 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Brief Fatigue Inventory change | 0-5 week
Brief Fatigue Inventory change | 6-11 week

SECONDARY OUTCOMES:
EORTC-QLQ-C30 change | 0-5 week, 6-11 week
EORTC-QLQ-BR23 change | 0-5 week, 6-11 week

CONTACTS AND LOCATIONS:
Locations (1):
- International St. Mary's Hospital, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cheon C, Kang S, Ko Y, Kim M, Jang BH, Shin YC, Ko SG. Sipjeondaebo-tang in patients with breast cancer with fatigue: a protocol for a pilot, randomised, double-blind, placebo-controlled, cross-over trial. BMJ Open. 2018 Jul 6;8(7):e021242. doi: 10.1136/bmjopen-2017-021242. PMID 29982213